CLINICAL TRIAL: NCT06617364
Title: Contrast Enhanced Multispectral Optoacoustic Tomography for Non-invasive Assessment of Intestinal Transit Time in Lactose Intolerance Patients
Brief Title: MSOT for Assessment of Intestinal Transit Time in Lactose Intolerance Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Ferdinand Knieling, PD Dr. med. Dr. rer. biol. hum., University Hospital Erlangen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MSOT_ICG_LI
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-11

CONDITIONS: Lactose Intolerance
Keywords: MSOT; lactose intolerance; pediatric; ICG; gastrointestinal transit
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pediatric patients with suspected lactose intolerance (Experimental): On the one hand the patients will undergo the hydrogen breath test and on the other their gastrointestinal transit time will be measured using MSOT and ICG contrast agent.
  Interventions: Procedure: gastrointestinal transit time measurement using MSOT and ICG contrast agent

INTERVENTIONS:
Procedure: gastrointestinal transit time measurement using MSOT and ICG contrast agent — The subject arrives at the clinic in the morning, fasting according to the preparation instructions from the Childrens Hospital Erlangen for the H2 breath test. Before taking the liquid containing lactose and ICG, the first measurement is performed using MSOT, followed by the H2 breath test. After the liquid to be detected is fully consumed, the second H2 breath test measurement, which only takes a few minutes, is conducted. According to the official guidelines of the Childrens Hospital Erlangen, the hydrogen concentration in the breath is measured at 30-minute intervals. During the 30-minute breaks, further MSOT measurements are carried out, also at 30-minute intervals. Each of these only takes about 10 minutes, they do not interfere with the H2 breath test measurement routine. After the ninth and final H2 breath test measurement a final MSOT examination is conducted. Afterwards participants are offered an optional MRI examination, which can be used to measure intestinal motility.

SUMMARY:
The study aims to investigate gastrointestinal transit using multispectral optoacoustic tomography (MSOT) in a prospective diagnostic study involving patients suspected of primary or secondary lactose intolerance. These patients exhibit varying clinical symptoms and different results from the hydrogen breath test (H2 breath test).

Lactose intolerance is caused by a deficiency in the enzyme lactase, which is responsible for breaking down lactose into glucose and galactose. Without this breakdown, lactose is fermented by colon bacteria, leading to symptoms such as bloating and diarrhea. The prevalence of lactose intolerance is increasing, especially among children, and the current diagnostic gold standard is the hydrogen breath test, which, while specific, has limitations in sensitivity.

MSOT could fill this diagnostic gap by non-invasively measuring intestinal transit time and providing a more objective assessment of the condition.

The study will compare MSOT results with H2 breath test outcomes, particularly focusing on patients with varying disease durations and activity levels.

Additionally, participants are offered an optional MRI examination, which can be used to measure intestinal motility. This helps to further quantify the results of the MSOT examination and discover new findings regarding the extent of the disease.

MSOT could improve the sensitivity of lactose intolerance diagnosis, differentiate it from other conditions, and offer insights into disease management over time.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the subject
* Written informed consent of the subject's legal guardian
* Suspicion or diagnosis of lactose intolerance
* Age 6 to 18 years

General Exclusion Criteria:

* Pregnancy
* Breastfeeding mothers
* Tattoo in the examination area
* Subcutaneous fat tissue over 3 cm
* Known hypersensitivity to ICG, sodium iodide, or iodine
* Hyperthyroidism, focal or diffuse thyroid autonomy
* Recent treatment for thyroid function assessment involving radioactive iodine (within two weeks before or after the study)
* Impaired renal function
* Use of the following medications: beta-blockers, anticonvulsants, cyclopropane, bisulfite compounds, haloperidol, heroin, meperidine, metamizole, methadone, morphine, nitrofurantoin, opium alkaloids, phenobarbital, phenylbutazone, probenecid, rifamycin, any injection containing sodium bisulfite

MRI Exclusion Criteria:

* General contraindications for MRI examinations (e.g., electrical implants such as pacemakers or infusion pumps, etc.)
* Severe claustrophobia

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
ICG-Signal in the intestinal tract | 1 day
  measured be MSOT

SECONDARY OUTCOMES:
Hydrogen breath test results | 1 day
  measured in ppm
MRI | 1 day
  peristaltic metrics

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Regensburger, PD Dr. med. Dr. rer. biol. hum, Study Chair
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No